CLINICAL TRIAL: NCT02527668
Title: To Test the Effect of Calcifediol Hy.D Supplementation on Muscle Function and Bone Quality in Younger Postmenopausal Women With Osteopenia: a Double-blind Randomized Placebo-controlled Trial
Brief Title: To Test the Effect of Calcifediol Hy.D Supplementation on Muscle Function and Bone Quality in Younger Postmenopausal Women With Osteopenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: University of Zurich (Other); Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2013-11-25-HyD-O; 000000198 (Other: SNCTP No.)
Record Dates: First submitted 2015-08-14; First posted 2015-08-19 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Osteopenia/Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Calcifediol; 25-hydroxyvitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Calcifediol Hy.D (25-hydroxyvitamin D) (Experimental): 20 μg Calcifediol Hy.D (25-hydroxyvitamin D) (one capsule) per day for 6 months
  Interventions: Dietary Supplement: Calcifediol
- Vitamin D3 (cholecalciferol) (Active Comparator): 3200 IU Vitamin D3 (cholecalciferol) (one capsule) per day for 6 months
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): 1 Placebo capsule per day for 6 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Calcifediol — One capsule orally of Calcifediol (20 µg) per day with a meal for a duration of 6 months
  Other Names: 25-hydroxyvitamin D (Hy.D)
  Arms: Calcifediol Hy.D (25-hydroxyvitamin D)
Dietary Supplement: Vitamin D3 — One capsule orally of Cholecalciferol (3200 IU) per day with a meal for a duration of 6 months
  Other Names: Cholecalciferol
  Arms: Vitamin D3 (cholecalciferol)
Other: Placebo — One capsule orally of a Placebo capsule per day with a meal for a duration of 6 months
  Arms: Placebo

SUMMARY:
Young postmenopausal women with osteopenia / or women with osteoporosis and a FRAX score below pharmacologic treatment indication have limited treatment options in the prevention of osteoporosis/treatment of osteopenia. Further, there is a concern about long-term side effects of bisphosphonate treatment among young postmenopausal women, and hormone replacement therapy has been controversial. In a pilot study 20 microgram Calcifediol Hy.D improved several muscle related function in this target population within 4 months of treatment, which can help to prevent falls and associated bone fractures. Thus the main aim of this study is to test whether Calcifediol Hy.D at a daily dose of 20 μg / day improves muscle function (lower extremity test battery) compared with (1) placebo and compared with (2) 3200 Vitamin D3 IU per day, at 3 and 6 month follow-up. As a secondary and exploratory objective of this study, the investigators will compare the beforementioned doses on muscle strength and the quality of the bones, beside muscle mass, body composition and systolic and diastolic blood pressure measurements.

ELIGIBILITY:
Inclusion Criteria:

* Women age 50 to 70
* Post-menopausal (defined as: at least 1 year after the last menstrual period)
* community-dwelling and ambulatory without help
* with documented osteopenia (BMD by DEXA t-score: < -1.0 and > -2.5 at the spine or hip) in the 6 months prior to enrolment or with documented osteoporosis (BMD by DEXA t-score: ≤ -2.5 at the spine or hip) and a FRAX score (online calculation tool of absolute 10 year fracture risk) below the Swiss age-dependent indication threshold for pharmacologic treatment for the 10-year risk of major osteoporotic fractures - at the screening visit and including DEXA (in the 6 months prior to enrolment) as part of the calculation
* body mass index > 18.5 and < 30 kg/m2
* 25(OH)D level < 24 µg/l (< 60 nmol/l)
* understands German in reading and writing plus able to read, understand, and complete questionnaires and tests
* willingness to limit additional vitamin D3 intake to 800 IU per day
* willingness to limit calcium supplement intake to 500 mg/day
* willingness to stop active vitamin D metabolites
* participant understands the study procedures, alternative treatments available and risks involved with the study and voluntarily agrees to participate by giving a written informed consent
* participant meets the routine clinical laboratory safety screening tests performed at screening visit
* participant is able and willing to perform all study tests, attend all required office visits, and provide blood and urine samples
* participant is able to swallow the study medication

Exclusion Criteria:

* Consumption of more than 1'000 IU vitamin D on any day in the 4 weeks prior to enrollment.
* Elevated serum calcium > 2.60 mmol/l adjusted for albumin if albumin ≤ 35 or ≥ 45g/l
* estimated creatinine clearance < 30 ml/min (Cockcroft and Gault = 140 - age(yr)*weight(kg)/ serum Cr(mmol/l))×(1.04 for women)
* severe visual or hearing impairment
* malabsorption syndrome (celiac diseases, inflammatory bowel disease).
* Pathologic fracture (excl. fractures due to osteoporosis) in the last year
* Fracture due to osteoporosis in the last 10 years
* Chemo therapy / Radiation due to cancer in the last year
* Treatment which has an effect on calcium metabolism (e.g. PTH, calcitonin, chronic cortisone intake > 5mg/day for more than 4 weeks in the last 12 months (except for inhalation and sporadic infiltration))
* Current treatment with a bisphosphonate
* For participants of the ancillary study "Muscle Biopsy" only: Treatment which has an effect on blood coagulation (e.g. factor X inhibitor, thrombin inhibitor, NSAR, low-molecular heparin, inhibitor for platelet aggregation, vitamin K antagonist) and/or abnormal blood coagulation status .
* Unwilling or unable to take study medication
* Diseases with a risk of recurrent falling (e.g. Parkinson's disease/syndrome, Hemiplegia after stroke, symptomatic stenosis of the spinal canal, polyneuropathy, epilepsy, recurring vertigo, recurring syncope)
* History of or current diseases that may enhance serum calcium: sarcoidosis, lymphoma, primary hyperparathyroidism
* Individual that heavily consumes alcohol containing products defined as greater than (>) 3 drinks (beer, wine, or distilled spirits) of alcoholic beverages per day.
* Individual is unlikely to adhere to the study procedures, to keep appointments, or is planning to relocate during the study.
* Individuals who are planning a stay in a "sunny" location (e.g. winter sun resort) for more than one month during the course of the study
* Medication which has an effect on 25-hydroxyvitamin D level (e.g. certain anticonvulsants (e.g. Phenobarbital, Carbamazepin, Phenytoin))
* M. Paget (Ostitis deformans)
* Inflammatory arthritis (e.g. rheumatoid arthritis, Reiter syndrome, psoriasis arthritis)
* Participation in a study in the last 6 months, except for studies without drug-application, or any influence of the study-medication can be excluded

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Overall assessment of the "lower extremity function" test battery (difference in proportion of those who improved or maintained function compared to those who declined in function by treatment group) | Baseline, 3 months, 6 months
  The "lower extremity function" test battery consists of: 8-meter walk test, repeated sit-to-stand test and knee flexion and extension strength test). A repeated measures analysis across all four test battery components simultaneously documenting the difference in proportion of those who improved or maintained function compared to those who declined in function by treatment group (comprised endpoint on lower extremity function) will be performed. Calcifediol Hy.D will be compared with (1) placebo and compared with (2) 3200 Vitamin D3 IU per day -for the time points baseline 3 and 6 months. Outcomes of the individual tests are subject to the secondary outcome measures.

SECONDARY OUTCOMES:
Gait speed measurement (8-meter walk) | Baseline, 3 months, 6 months
Knee flexion and extension strength test | Baseline, 3 months, 6 months
Repeated sit-to-stand test (reaction time) | Baseline, 3 months, 6 months
Systolic and diastolic blood pressure | Baseline, 3 months, 6 months
Timed up and go test (functional mobility) | Baseline, 3 months, 6 months

OTHER OUTCOMES:
Bone mineral density (DXA) | Baseline and 6 months
  spine, hip (both sides at baseline, side with lowest total femur BMD only at follow-up), radius
Muscle mass (DXA) | Baseline and 6 months
  Upper and lower extremity, body composition
Bone quality (Xtreme CT): | Baseline and 6 months
  Tibia (funding is pending), radius (funding is pending)
Cognition (MoCa test score) | Baseline and 6 months
  MoCa: Montreal Cognitive Assessment
Quality of life questionnaire | Baseline, 3 months, 6 months
  EuroQol country specific TTM Index
Upper extremity test (grip strength) | Baseline, 3 months, 6 months
Cardiovascular fitness (6-minute walking test) | Baseline, 3 months, 6 months
Cardio vascular risk marker (NT-BNP) | Baseline, 3 months, 6 months
Bone marker: P1NP | Baseline, 3 months, 6 months
Bone marker: Osteocalcin | Baseline, 3 months, 6 months
Bone marker: Sclerostin | Baseline, 3 months, 6 months
Muscle marker: myostatin | Baseline, 3 months, 6 months
Safety: Serum calcium adjusted for albumin | Screening, 3 months, 6 months
Safety: Serum creatinine | Screening, 3 months, 6 months
Safety: Urinary calcium/creatinine Ratio | Screening, 3 months, 6 months
Safety: Blood pressure | Screening, 3 months, 6 months
Safety: Pulse rate | Screening, 3 months, 6 months
Ancillary studies: Analysis of expression of the vitamin D receptor (VDR) in skeletal muscle | Baseline, 6 months
  18 of 50 participants in active group I, active group II and control will be enrolled in the muscle biopsy ancillary study. The muscle biopsies (about 0.2 g) will be taken from mid-thigh at baseline and at 6 months follow-up. Biopsies will be taken at the Zurich site, frozen and send to the Tufts University Boston, USA for analysis. Analysis: Expression of the vitamin D receptor (VDR) in skeletal muscle
Ancillary studies: Analysis of total cross-sectional area (CSA) of muscle fibers | Baseline, 6 months
  18 of 50 participants in active group I, active group II and control will be enrolled in the muscle biopsy ancillary study. The muscle biopsies (about 0.2 g) will be taken from mid-thigh at baseline and at 6 months follow-up. Biopsies will be taken at the Zurich site, frozen and send to the Tufts University Boston, USA for analysis. Analysis: Total cross-sectional area (CSA) of muscle fibers
Ancillary studies: Dried blood spot | Baseline, 3 months
  Among all 150 participants, we compare 25(OH)D content in arterial finger tip blood and venous blood at baseline and at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Heike Bischoff-Ferrari, Prof, Dr.PH, Principal Investigator — Center on Aging and Mobility, Klinik für Geriatrie, UniversitätsSpital Zürich
Locations (1):
- Center on Aging and Mobility, Klinik für Geriatrie, UniversitätsSpital Zürich, Zurich, Switzerland

REFERENCES:
- [Derived] Bischoff-Ferrari HA, Dawson-Hughes B, Orav JE, Ceglia L, Egli A, Kistler-Fischbacher M, Wieczorek M, de Godoi Rezende Costa Molino C. Effect of calcifediol and cholecalciferol on muscle function in postmenopausal women: a randomized controlled trial. Osteoporos Int. 2025 Jun;36(6):1007-1018. doi: 10.1007/s00198-025-07456-7. Epub 2025 Apr 9. PMID 40205202
- [Derived] Ceglia L, Rivas DA, Schlogl M, Fielding GB, Egli A, Bischoff-Ferrari HA, Dawson-Hughes B. Effect of vitamin D3 vs. calcifediol on VDR concentration and fiber size in skeletal muscle. J Bone Miner Metab. 2023 Jan;41(1):41-51. doi: 10.1007/s00774-022-01374-y. Epub 2022 Nov 16. PMID 36385193